CLINICAL TRIAL: NCT04039490
Title: Novel Device for Ultrasound-guided Pediatric Vessel Cannulations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clear Guide Medical (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); Children's National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CNMC Ph II Trial
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Clinical Procedures Which Require Vessel Cannulations in Pediatric Patients
Keywords: pediatrics; vessel cannulations; ultrasound-guided

STUDY DESIGN:
Intervention Model Description: two-arm study, comparing ultrasound-only pediatric vessel cannulations versus SCENERGY-guided pediatric vessel cannulations
Masking Description: Because the SCENERGY is an attachment to the ultrasound probe, it cannot be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Ultrasound-only Pediatric Vessel Cannulation (No Intervention): The standard of care for vessel cannulation currently employed at CNMC
- SCENERGY-guided Pediatric Vessel Cannulation (Experimental): The addition of the SCENERGY guidance combined with the ultrasound for pediatric vessel cannulations.
  Interventions: Device: SCENERGY

INTERVENTIONS:
Device: SCENERGY — Use of the SCENERGY guidance device in conjunction with ultrasound to guide needles for pediatric vessel cannulations
  Arms: SCENERGY-guided Pediatric Vessel Cannulation

SUMMARY:
Clinical Trial to investigate whether the use of a novel device to be used in conjunction with ultrasound in pediatric vessel cannulations is superior to ultrasound-only pediatric vessel cannulations in terms of number of cannulation attempts.

DETAILED DESCRIPTION:
Use of needle guidance plus ultrasound imaging for CVC placement in the pediatric high-risk population may facilitate the procedure with a single needle pass and decrease the incidence of adverse effects by minimizing additional needle passes. This study will compare the use of ultrasound-only guidance with the Clear Guide SCENERGY guidance in terms of successful first-attempt vessel cannulations such as internal jugular and fermoral artery access. The question is whether it is possible to make ultrasound-guided pediatric vascular access less technically challenging in order to improve adoption and utilization leading to decreased iatrogenic complications and improved patient safety.

ELIGIBILITY:
Inclusion Criteria:

* any pediatric patient scheduled for a vessel cannulation at CNMC

Exclusion Criteria:

* none

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Successful first-attempt vessel cannulation | 1 hour
  Test if the vessel cannulation was successful with only 1 attempt --needle puncture--to reach the vessel

SECONDARY OUTCOMES:
Non-IR Personnel Successfully Cannulate Pediatric Patients | 1 hour
  Test if non-specialists can learn to successfully cannulate pediatric patients with only 1 needle puncture.
Point-of-Care Successful Cannulation | 1 hour
  Test whether the SCENERGY makes possible successful pediatric vessel cannulations at patient's point of care location.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No